CLINICAL TRIAL: NCT05347433
Title: Comparison of 18-24 Week Pregnant Women With in Vitro Fertilization (IVF) and Pregnant Women With Spontaneous Pregnancy in the Same Week in Terms of Fetal Thymus Volume
Brief Title: Comparison of Fetal Thymus Volumes of Pregnant Women With In Vitro Fertilization (IVF) and Spontaneous Pregnant Women.
Status: Completed | Type: Observational
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Nurgül Selin KAYA, doctor, Karadeniz Technical University
Other Study IDs: 2019/205
Record Dates: First submitted 2022-04-21; First posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Healthy
Keywords: Fetal thymus volume; In vitro fertilization

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tube baby pregnancy group: 18-24-week pregnant women with in vitro fertilization
- Spontaneous pregnancy group: 18-24-week pregnant women with spontaneous

SUMMARY:
The purpose of the study was to compare the fetal thymus volumes of 18-24-week pregnant women with In Vitro Fertilization (IVF) and spontaneous pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* pregnant between 18-24 weeks
* had no complaints
* between the ages of 18-35
* conceived with in vitro fertilization or spontaneously

Exclusion Criteria:

* history of endocrinopathies (including diabetes mellitus, hyperprolactinemia, Cushing's disease, and congenital adrenal hyperplasia), systemic diseases (e.g. asthma), collagen disorder, hypercholesterolemia, sickle cell anemia, or neoplasm,
* those who had a history of coronary artery disease, angina, or myocardial infarction, or a history of hypertension, coronary arteritis, and electrocardiographic changes that suggest any known history of vascular, infectious, or inflammatory disease, maternal autoimmune disease,
* use of any drugs other than those used for IVF (e.g. insulin sensitizing drugs, oral contraceptives, antiandrogens, statins, aspirin, and corticosteroids) in the 3 months before the pregnancy,
* multiple pregnancy,
* present cigarette and alcohol use,
* abnormal renal, hepatic, and thyroid function test results;
* refusing to participate in the study,
* abnormal fetal findings (fetal anomaly, increased nape transparency, first-second trimester screening test disorder),
* cases who did not meet the criteria for pregnancy after the first tube treatment (ICSI-ET) because of normoresponder, unexplained infertility, or male factor

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study group consisted of normal pregnant women who applied to the pregnancy clinic for routine pregnancy follow-ups
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2019-07-09 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
measurement of fetal thymus volume | 18-24 week pregnant women
  The thymus is located at the superior part of the fetal rib cage. When the transverse section, which includes three vessel images (Superior Vena Cava, Aorta, Pulmonary Artery) is taken, fetal sternum is observed between the three-vessel view and fetal lungs. It is found as a hypoechoic two-lobe structure in the anterior mediastinum compared to other tissues. The fetal thymus dimensions were evaluated by one single person by using the VOLUSON E-10 ultrasonography, which can make VOCAL measurements with 2D and 3D VOCAL Program in 3-vessel trachea sections.

SECONDARY OUTCOMES:
frequency of pregnancy complications | during pregnancy and at delivery week
  The cases were followed up during pregnancy and at delivery week, and frequency of preeclampsia, non-reliable fetal status, Intrauterine growth restriction and neonatal intensive care requirement wererecorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Karadeniz Technical University, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided